CLINICAL TRIAL: NCT06171620
Title: Virtual Reality as a Non-pharmacological Tool for Pain and Anxiety Relief During Elective Procedures in the Cathlab
Brief Title: Virtual Sedation During Elective Procedures in the Cathlab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22283VR Cathlab
Record Dates: First submitted 2023-09-08; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two group design, Standard of care (control) vs Standard of care + VR intervention (Intervention group)
Masking Description: Due to the visual presence of the VR, masking is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (SOC) (Other): Standard of care
  Interventions: Other: Standard of care
- Intervention Group (VR) (Experimental): Standard of care with addition of the Virtual reality headset
  Interventions: Device: Virtual reality headset

INTERVENTIONS:
Device: Virtual reality headset — Distraction therapy using a virtual reality headset. Participants will access a digitally created environment such as a forest or sub sea exploration with relaxing auditory cues.
  Arms: Intervention Group (VR)
Other: Standard of care — Elective procedure performed as planned according to current standard of care in the hospital.
  Arms: Control group (SOC)

SUMMARY:
This study aims to investigate the effectiveness of virtual reality (VR) as a non-pharmacological tool against anxiety and pain during elective procedures in the catheterization laboratory (cathlab).

To assess the effectiveness of VR in the clinical setting of daily practice within the cathlab, a comparative effectiveness trial will be conducted. A sample of patients scheduled for a planned procedure in the cathlab of UZ Brussel will be selected using convenience sampling.

Participants eligible for this study will be assigned to either the control group or the intervention group after signing the informed consent form. The control group in this study will receive standard care according to current practice for the planned procedure, while the intervention group will receive standard care along with the virtual reality headset intervention.

The primary outcome of anxiety will be measured using the Visual Analog Scale (VAS) for anxiety and the State-Trait Anxiety Inventory (STAI) questionnaire. The secondary outcome of pain will be measured using the VAS scale for pain.

Other outcomes such as satisfaction and potential nausea during the procedure will be assessed through a questionnaire that participants will fill out after the procedure. The physician who performed the procedure in the intervention group, as well as the involved nurses during the procedure, will complete a similar questionnaire to evaluate the use of the VR headset from the operators' perspective.

The outcomes of the two groups will be statistically compared using the SPSS software package.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective procedure in line with the following criteria in the cathlab of the UZB: limited feedback requirements from the patient to the physician, per-formed under local anaesthesia, risk estimated as normal i.e. haemodynamically stable patients (Stable vital signs such as heart rate and blood pressure) and no expected complications, electively planned and duration expected to be between 30 minutes and two hours.
* Agreeing to participate via signed informed consent.
* Being at least 18 years of age.
* Being fluent in either English, French or Dutch language.

Exclusion Criteria:

* Ailments which would make wearing of the headset uncomfortable or impossible.
* cognitive impairment such as dementia or delirium.
* Severe hearing impairment, as this will limit the immersion.
* Severe visual impairment not compensated by glasses, such as blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Anxiety | State trait: 30 minutes pre operatively and 5 minutes post operatively. Anxiety using VAS: 5 min pre operatively for baseline and 5 minutes post operatively.
  perioperative anxiety consisting of State, trait anxiety and anxiety experienced during the procedure.
  State anxiety: level of anxiety a person experiences in the current moment. Trait anxiety: Level of anxiety a person experiences in general, how anxious a person is in general.
  State and trait anxiety will be measured using the state trait anxiety inventory questionnaire consisting of 20 questions for state anxiety and 20 questions for trait anxiety. The questions are answered in the form of Likert scales ranging from 1 to 4.
  Anxiety experienced during the procedure will be measured using the visual analogue scale (VAS) which ranges from 0 (none) to 100 mm (worst imaginable).
Pain experienced during the procedure | using VAS: 5 min pre operatively for baseline and 5 minutes post operatively.
  The level of pain a patient experienced throughout the elective procedure measured using the Visual analogue scale (VAS) which ranges from 0 (none) to 100 mm (worst imaginable).

SECONDARY OUTCOMES:
Procedural comfort | 5 minutes after the procedure
  Patient experience during the elective procedure. This will be assessed by a custom patient questionnaire with the question: how was your experience during the procedure? The answer will be in the form of a scale ranging from 1 (very uncomfortable) to 10 (very comfortable).
  This questionnaire will be given to the patient 5 minutes after the end of the procedure.
Operator comfort (nurses and doctors). | 5 minutes after the procedure.
  How the nurses and doctors experienced the procedure and level of support they needed to provide the patient.
  This will be assessed by a custom questionnaire with the question: To what degree did you need to provide reassurance to the patient during this procedure? The answer will be in the form of a Likert scale ranging from 1 (No reassurance needed) to 5 (Continuous reassurance needed).
  This questionnaire will be given to the patient 5 minutes after the end of the procedure.
Nausea | 5 minutes after the procedure
  The level of nausea (If any) a patient experienced during the procedure. This will be assessed by a custom questionnaire with the question: to what degree did you experience nausea during this procedure? The answer will be in the form of a scale ranging from 0 (none) to 10 (severe).
  This questionnaire will be given to the patient 5 minutes after the end of the procedure.
Systolic blood pressure | At the start of the procedure and every 15 minutes.
  The systolic blood pressure will be measured none invasively every 15 minutes during the procedure using the M540 infinity monitoring system by Dräger.
Diastolic blood pressure | At the start of the procedure and every 15 minutes.
  The Diastolic blood pressure will be measured none invasively every 15 minutes during the procedure using the M540 infinity monitoring system by Dräger.
Mean Blood pressure | At the start of the procedure and every 15 minutes.
  The mean blood pressure will be measured none invasively every 15 minutes during the procedure using the M540 infinity monitoring system by Dräger.
Heart rate | At the start of the procedure and every 15 minutes.
  Heart rate will be measured every 15 minutes alongside the NIBP. This will be done by using both the pulse oximetry device and ECG monitoring system from Philips.
Satisfaction with VR (for patient, nurses and doctors) | 5 minutes after the procedure
  Satisfaction with VR will be assessed by a custom questionnaire with the following questions:
  * Was the VR headset an added value for you during this procedure?
  * To which degree would you recommend the use of the VR headset during this procedure?
  These questions are answered by Likert scales ranging from 1 (none at all) to 5 (greatly so).
  The questionnaires include several open ended questions for potential problems that occurred due to the presence of the VR headset and any personal remarks.

CONTACTS AND LOCATIONS:
Overall Officials: Johan De Sutter, PHD, MD, Principal Investigator — University Ghent
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No